CLINICAL TRIAL: NCT02293369
Title: Comparison of Two Methods of Vaginal Cuff Closure at Laparoscopic Hysterectomy and Their Effect on Female Sexual Function and Vaginal Length
Brief Title: Comparison of Two Methods of Vaginal Cuff Closure at Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Principal Investigator, Ercan Bastu, Associate Professor of Obstetrics and Gynecology, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1424
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Total Laparoscopic Hysterectomy; Benign Conditions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cuff closure via vaginal route (Active Comparator): For vaginal cuff closure both in laparoscopic approach and vaginal route, we will use the same horizontal method, which can be described as closing the vagina anterior to posterior by leaving a horizontal scar. The repair will start at one end of the vaginal cuff, taking care to incorporate the uterosacral ligament into the initial bite and will continue toward the surgeon until the other uterosacral ligament will be incorporated into the repair, using a continuous 0-Vicryl suture in the vaginal route.
  Interventions: Procedure: Cuff closure via vaginal route
- Cuff closure via laparoscopic route (Active Comparator): For vaginal cuff closure both in laparoscopic approach and vaginal route, we will use the same horizontal method, which can be described as closing the vagina anterior to posterior by leaving a horizontal scar. In the laparoscopic approach, needles will be introduced through the umbilical trocar and removed through the peripheral trocars and intracorporeal knots will be utilized.
  Interventions: Procedure: Cuff closure via laparoscopic route

INTERVENTIONS:
Procedure: Cuff closure via vaginal route — Vaginal cuff will be closed via vaginal route during total laparoscopic hysterectomy.
  Arms: Cuff closure via vaginal route
Procedure: Cuff closure via laparoscopic route — Vaginal cuff will be closed via laparoscopic route during total laparoscopic hysterectomy.
  Arms: Cuff closure via laparoscopic route

SUMMARY:
American Congress of Obstetricians and Gynecologists (ACOG) advises minimally invasive methods in gynecological surgery to ensure increased benefits to the patient and reduce potential hospitalization costs.

Laparoscopic hysterectomy has become the standard approach in gynecological benign disorders. During laparoscopic hysterectomy, vaginal cuff can be closed with different sutures, techniques and approaches, which is one of the challenges of this surgery. Data is limited on potential impact of different sutures, techniques and approaches for vaginal cuff closure on female sexual function in relation to vaginal length.

Various studies in the literature evaluated different approaches (abdominal, vaginal, laparoscopic, robotic-assisted laparoscopic). In addition, for cuff closure, different techniques (interrupted, continuous) and sutures (barbed, Vicryl) were compared. Measures like operation time, cuff healing, complications, cost effectiveness, etc. were usually measured. However, there is no prospective randomized clinical study in the literature that compares laparoscopic approach with vaginal route for cuff closure in terms of female sexual function in relation to vaginal length.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have total laparoscopic hysterectomy because of benign conditions only

Exclusion Criteria:

* Suspicion of malignancy
* Presence of large adnexal masses (maximum diameter >10 cm at preoperative ultrasonography)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function | Three months
  Patients will be asked to fill out female sexual function index (FSFI) prior to surgery and at the 3-month follow-up.
Vaginal length | One months
  Vaginal measure will be taken prior to surgery and at 1-month follow-up.

SECONDARY OUTCOMES:
Vaginal cuff granulation/infection | One month
  Vaginal cuff granulation and any evidence of vaginal cuff infection will be carefully examined and documented during the 4-week follow-up visit
Vaginal cuff closure time | One day
  Cuff closure time will be recorded for each patient during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Buyru, M.D., Study Chair — Istanbul University School of Medicine
Locations (1):
- Department of Obstetrics and Gynecology, Istanbul University School of Medicine, Istanbul, Turkey (Türkiye)